CLINICAL TRIAL: NCT04871555
Title: Structural Cartography of the Insula in Temporal Epilepsy Patients
Acronym: CON-INSULA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); University Hospital, Lille (Other); Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, TYVAERT Louise, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI218
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Epilepsy, Temporal Lobe; MRI Scans
Keywords: structural connectivity; insula; temporal lobe epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- mesio-temporal epilepsy: patients suffering from mesiotemporal epilepsy type
  Interventions: Other: MRI
- basal temporal epilepsy: patients suffering from basal temporal epilepsy type
  Interventions: Other: MRI
- temporal lateral epilepsy: patients suffering from temporal lateral epilepsy type
  Interventions: Other: MRI
- operculo insular epilepsy: patients suffering from operculo insular epilepsy type
  Interventions: Other: MRI
- temporo-insular epilepsy: patients suffering from temporo- insular epilepsy type
  Interventions: Other: MRI
- healthy subjects: non epileptic patients
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — structural imaging

SUMMARY:
The purpose of this study is to investigate insula structural connectivity in temporal epilepsy patients. Insula being at the interface of frontal, parietal, occipital and temporal lobes, its structural organization reflects the brain function. We hypothetize that insular structural organization will be different according to the different subtypes of temporal epilepsy.

DETAILED DESCRIPTION:
The purpose of this study is to investigate insula structural connectivity in temporal epilepsy patients. Insula being at the interface of frontal, parietal, occipital and temporal lobes, its structural organization reflects the brain function. We hypothetize that insular structural organization will be different according to the different subtypes of temporal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* epileptic patients: temporal epilepsy or temporal plus epilepsy (temporomesial epilepsy, basal temporal epilepsy, mesio lateral or lateral epilepsy, temporo insular epilepsy, operculo insular epilepsy)
* patients who underwent video EEG monitoring with recorded seizures (at least one)
* patients who underwent a brain MRI with DTI sequence before epilepsy surgery
* patients who did not refuse the use of their clinical and MRI data for this study

Exclusion Criteria:

* patients younger than 15 years old
* patients with previous brain surgery (before MRI)
* uncompleted MRI sequences (DTI, T1 anatomical)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: temporal epilepsy patients and healthy subjects
  healthy subjects will be selected in the healthy cohort of Nguyen G-Dang (Ghaziri et al., 2017)
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
cartography of insula in temporal epilepsy patients | 1 year after the last inclusion
  Compared with healthy group, definition of different patterns of insular structural connectivity in epileptic patients

SECONDARY OUTCOMES:
Correlation structural cartography and electroclinical data | 1 year after the last inclusion
  correlation between patterns of insular structural connectivity and subtypes of epilepsy defined by electroclinical data

CONTACTS AND LOCATIONS:
Overall Officials: Louise Tyvaert, MD PHD, Principal Investigator — CHRU Nancy, CRAN UMR 7039 Université de Lorraine
Locations (1):
- Central Hospital nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No